CLINICAL TRIAL: NCT02317705
Title: A Phase 2, Single Dose, Open-Label Study to Investigate the Safety and Efficacy of OTL38 Injection (OTL38) for Intra-operative Imaging of Folate Receptor-alpha Positive Ovarian Cancer
Brief Title: Phase 2 Study of OTL38 for Intra-operative Imaging of Folate Receptor-alpha Positive Ovarian Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: On Target Laboratories, LLC (Industry)
Collaborators: SynteractHCR (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: OTL-2014-OTL38-003
Record Dates: First submitted 2014-11-18; First posted 2014-12-16 (Estimated); Results first posted 2022-06-21 (Actual); Last update posted 2022-06-21 (Actual); Status verified 2022-05

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Pafolacianine; Injections; Laparotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Patients Receiving OTL38 (Experimental): All patients in this arm will receive OTL38 for injection and undergo intraoperative imaging.
  Interventions: Drug: OTL38; Device: Near infrared camera imaging system; Procedure: Laparotomy

INTERVENTIONS:
Drug: OTL38
  Other Names: OTL38 for Injection; CYTALUX™ (pafolacianine) injection
Device: Near infrared camera imaging system — Near infrared camera imaging system
Procedure: Laparotomy — primary surgical cytoreduction, interval debulking, or recurrent ovarian cancer surgery

SUMMARY:
This study is being done to:

* test the safety of OTL38
* see if OTL38 helps light up the cancer when viewed with the special camera system
* test the safety of the special camera system for use along with OTL38 during surgery

ELIGIBILITY:
Inclusion Criteria:

1. Female patients 18 years of age and older
2. Have a primary diagnosis, or at high clinical suspicion, of primary ovarian cancer (of epithelial type), planned for primary debulking or interval debulking surgery, and:

   * Who are scheduled to undergo laparotomy for the debulking surgery OR
   * Who are scheduled to undergo laparoscopy and pre-authorized to undergo laparotomy for the debulking surgery, if cancer is detected on the laparoscopy
3. A negative serum pregnancy test at Screening followed by a negative urine pregnancy test on the day of surgery or day of admission for female patients of childbearing potential
4. Female patients of childbearing potential or less than 2 years postmenopausal agree to use an acceptable form of contraception from the time of signing informed consent until 30 days after study completion
5. Ability to understand the requirements of the study, provide written informed consent and authorization of use and disclosure of protected health information, and agree to abide by the study restrictions and to return for the required assessments

Exclusion Criteria:

1. Previous exposure to OTL38
2. Known FR alpha-negative ovarian cancer
3. Planned surgical approach via laparoscopy or robotic surgery
4. Any medical condition that in the opinion of the investigators could potentially jeopardize the safety of the patient
5. History of anaphylactic reactions or severe allergies
6. History of allergy to any of the components of OTL38, including folic acid
7. Pregnancy, or positive pregnancy test
8. Clinically significant abnormalities on electrocardiogram (ECG)
9. Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule
10. Impaired renal function defined as eGFR< 50 mL/min/1.73m2
11. Impaired liver function defined as values > 3x the upper limit of normal (ULN) for alanine aminotransferase (ALT) or aspartate aminotransferase (AST), alkaline phosphatase (ALP), or total bilirubin.
12. Known Stage IV ovarian cancer with Brain Metastases
13. Received an investigational agent in another investigational drug or vaccine trial within 30 days prior to surgery
14. Known sensitivity to fluorescent light

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2014-12; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - University of CA at Irvine Chao Cancer Center, Orange, California
  - Moffitt Cancer Center, Tampa, Florida
  - Mayo Clinic-Rochester, Rochester, Minnesota
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Al Rawahi T, Lopes AD, Bristow RE, Bryant A, Elattar A, Chattopadhyay S, Galaal K. Surgical cytoreduction for recurrent epithelial ovarian cancer. Cochrane Database Syst Rev. 2013 Feb 28;2013(2):CD008765. doi: 10.1002/14651858.CD008765.pub3. PMID 23450588
- [Background] Crane LM, Arts HJ, van Oosten M, Low PS, van der Zee AG, van Dam GM, Bart J. The effect of chemotherapy on expression of folate receptor-alpha in ovarian cancer. Cell Oncol (Dordr). 2012 Feb;35(1):9-18. doi: 10.1007/s13402-011-0052-6. Epub 2011 Jun 7. PMID 21647742
- [Background] Ibeanu OA, Bristow RE. Predicting the outcome of cytoreductive surgery for advanced ovarian cancer: a review. Int J Gynecol Cancer. 2010 Jan;20 Suppl 1:S1-11. doi: 10.1111/IGC.0b013e3181cff38b. PMID 20065732
- [Background] Kalli KR, Oberg AL, Keeney GL, Christianson TJ, Low PS, Knutson KL, Hartmann LC. Folate receptor alpha as a tumor target in epithelial ovarian cancer. Gynecol Oncol. 2008 Mar;108(3):619-26. doi: 10.1016/j.ygyno.2007.11.020. Epub 2008 Jan 28. PMID 18222534
- [Background] Leamon CP, Low PS. Membrane folate-binding proteins are responsible for folate-protein conjugate endocytosis into cultured cells. Biochem J. 1993 May 1;291 ( Pt 3)(Pt 3):855-60. doi: 10.1042/bj2910855. PMID 8387781
- [Background] Markert S, Lassmann S, Gabriel B, Klar M, Werner M, Gitsch G, Kratz F, Hasenburg A. Alpha-folate receptor expression in epithelial ovarian carcinoma and non-neoplastic ovarian tissue. Anticancer Res. 2008 Nov-Dec;28(6A):3567-72. PMID 19189636
- [Background] Parker N, Turk MJ, Westrick E, Lewis JD, Low PS, Leamon CP. Folate receptor expression in carcinomas and normal tissues determined by a quantitative radioligand binding assay. Anal Biochem. 2005 Mar 15;338(2):284-93. doi: 10.1016/j.ab.2004.12.026. PMID 15745749
- [Background] Ross JF, Chaudhuri PK, Ratnam M. Differential regulation of folate receptor isoforms in normal and malignant tissues in vivo and in established cell lines. Physiologic and clinical implications. Cancer. 1994 May 1;73(9):2432-43. doi: 10.1002/1097-0142(19940501)73:93.0.co;2-s. PMID 7513252
- [Background] Shih KK, Chi DS. Maximal cytoreductive effort in epithelial ovarian cancer surgery. J Gynecol Oncol. 2010 Jun;21(2):75-80. doi: 10.3802/jgo.2010.21.2.75. Epub 2010 Jun 30. PMID 20613895
- [Background] Toffoli G, Russo A, Gallo A, Cernigoi C, Miotti S, Sorio R, Tumolo S, Boiocchi M. Expression of folate binding protein as a prognostic factor for response to platinum-containing chemotherapy and survival in human ovarian cancer. Int J Cancer. 1998 Apr 17;79(2):121-6. doi: 10.1002/(sici)1097-0215(19980417)79:23.0.co;2-v. PMID 9583724
- [Background] van Dam GM, Themelis G, Crane LM, Harlaar NJ, Pleijhuis RG, Kelder W, Sarantopoulos A, de Jong JS, Arts HJ, van der Zee AG, Bart J, Low PS, Ntziachristos V. Intraoperative tumor-specific fluorescence imaging in ovarian cancer by folate receptor-alpha targeting: first in-human results. Nat Med. 2011 Sep 18;17(10):1315-9. doi: 10.1038/nm.2472. PMID 21926976
- [Background] Weitman SD, Lark RH, Coney LR, Fort DW, Frasca V, Zurawski VR Jr, Kamen BA. Distribution of the folate receptor GP38 in normal and malignant cell lines and tissues. Cancer Res. 1992 Jun 15;52(12):3396-401. PMID 1596899

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Subjects were screened up to 28 days prior to surgery.
Groups:
- OTL38 for Intra-operativeImaging of Folate Receptor-alpha Positive Ovarian Cancer: Patient injected with a dose of 0.025 mg/kg OTL38 and undergoes intraoperative imaging
Period: Overall Study
Arm/Group | OTL38 for Intra-operativeImaging of Folate Receptor-alpha Positive Ovarian Cancer
Started | 48
Safety Population (All patients who received OTL38.) | 44
Modified Intent-to-Treat (mITT) (All patients who received OTL38, underwent cytoreductive surgery, were exposed to fluorescent light using the imaging system, and had at least one Folate Receptor-alpha positive target ovarian cancer lesion. Patients enrolled after protocol amendment 4 will not be included in the mITT population.) | 29
Completed (Four subjects were screen failures and did not receive treatment; one subject who received treatment did not complete the study) | 43
Not Completed | 5
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Not completed — Drug not usable | 1

BASELINE CHARACTERISTICS:
Population: Number of enrolled subjects
Groups:
- OTL38 for Intra-operative Imaging of Folate Receptor-alpha Positive Ovarian Cancer: Patient injected with a dose of 0.025 mg/kg OTL38 and undergoes intraoperative imaging
Arm/Group | OTL38 for Intra-operative Imaging of Folate Receptor-alpha Positive Ovarian Cancer
Number analyzed (Participants) | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 21
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.8 (10.19)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 37
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 35
  More than one race | 1
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United States | 44

OUTCOME MEASURES:

1. Primary Outcome: Sensitivity of OTL38 in Detecting Folate Receptor-alpha Positive Ovarian Cancer During Surgery.
Description: Sensitivity for the detection of folate receptor-alpha positive (FRAP) ovarian cancer lesions is defined as the ratio (multiplied by 100) of the number of FRAO ovarian cancer lesions confirmed by both fluorescent light and the pathology/ and immunohistochemistry lab (TP) over the number of FRAP ovarian cancer lesions confirmed by the pathology/ and immunohistochemistry lab (TP+FN). 95% lower one-sided confidence interval was used.
Time Frame: Day of Surgery (Day 1)
Population: Population includes all patients who received OTL38, underwent cytoreductive surgery for sensitivity analysis, were exposed to fluorescent light using the imaging system, and had at least one FRAP target ovarian cancer lesion. Patients enrolled to the study after adequate number of lesions have been excised and submitted for pathology, and immunohistochemistry evaluation for determining sensitivity, enrolled after protocol amendment 4, were not included in the analysis population.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions
Groups:
- Experimental: Patient injected with a dose of 0.025 mg/kg OTL38 and undergoes intraoperative imaging
Arm/Group | Experimental
Number analyzed (Participants) | 29
Number analyzed (lesions) | 225
percentage of lesions | 97.97 [87.75 to NA] — data are not available to report the upper limit as the 95% lower one sided Confidence Interval is calculated according to the pre-specified analysis plan

2. Primary Outcome: Positive Predictive Value (PPV) of OTL38 in Detecting Folate Receptor-alpha Positive Ovarian Cancer During Surgery.
Description: PPV for the detection of FRAP ovarian cancer lesions is defined as the ratio (multiplied by 100) of the number of FRAP ovarian cancer lesions confirmed by both fluorescent light and the pathology/ and immunohistochemistry lab (TP) over the number of FRAP ovarian cancer lesions confirmed by fluorescent light (TP + FP).
  95% lower one-sided confidence interval was used.
Time Frame: Day of Surgery (Day 1)
Population: Population includes all patients who received OTL38, underwent cytoreductive surgery for PPV analysis, were exposed to fluorescent light using the imaging system, and had at least one FRAP target ovarian cancer lesion. Patients enrolled to the study after adequate number of lesions have been excised and submitted for pathology, and immunohistochemistry evaluation for determining PPV, enrolled after protocol amendment 4, were not included in the analysis population.
Measure: Number (95% Confidence Interval); unit: percentage of lesions
Units Other Than Participants: lesions
Arm/Group | Experimental
Number analyzed (Participants) | 29
Number analyzed (lesions) | 225
percentage of lesions | 94.93 [86.13 to NA] — data are not available to report the upper limit as the 95% lower one sided Confidence Interval is calculated according to the pre-specified analysis plan

ADVERSE EVENTS:
Time Frame: Adverse events were collected from the time of study drug administration throughout the course of the study, ending with Visit 4. The total collection period for each subject was approximately one month.
Description: The definition of AEs and SAEs for this study was consistent with the clinicaltrials.gov definitions.
Groups:
- Patients Receiving OTL38: All patients in this arm will receive OTL38 for injection and undergo intraoperative imaging.
  OTL38
  Near infrared camera imaging system: Near infrared camera imaging system
  Laparotomy: primary surgical cytoreduction, interval debulking, or recurrent ovarian cancer surgery
Arm/Group | Patients Receiving OTL38
All-Cause Mortality (participants affected / at risk) | 0/44
Serious Adverse Events (participants affected / at risk) | 13/44
Other Adverse Events (participants affected / at risk) | 44/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Receiving OTL38 (N=44)
Postoperative wound infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Septic Shock (Infections and infestations) | 1 (1)
Wound abscess (Infections and infestations) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Plueral effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 1 (1)
Haematoma (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 1 (1)
Pyrexia (General disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Patients Receiving OTL38 (N=44)
Nausea (Gastrointestinal disorders) | 12 (14)
Vomiting (Gastrointestinal disorders) | 14 (14)
Abdominal distension (Gastrointestinal disorders) | 4 (5)
Constipation (Gastrointestinal disorders) | 4 (5)
Diarrhoea (Gastrointestinal disorders) | 4 (4)
Dysphagia (Gastrointestinal disorders) | 3 (3)
Ileus (Gastrointestinal disorders) | 3 (3)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Ascites (Gastrointestinal disorders) | 2 (2)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1)
Ileus paralytic (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Procedural pain (Injury, poisoning and procedural complications) | 40 (40)
Infusion related reaction (Injury, poisoning and procedural complications) | 5 (6)
Procedural nausea (Injury, poisoning and procedural complications) | 3 (3)
Bladder injury (Injury, poisoning and procedural complications) | 1 (1)
Gastrointestinal anastomotic leak (Injury, poisoning and procedural complications) | 1 (1)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 11 (15)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2)
Thrombocytosis (Blood and lymphatic system disorders) | 1 (1)
Urinary tract infection (Infections and infestations) | 3 (3)
Pneumonia (Infections and infestations) | 2 (2)
Postoperative wound infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Clostridium difficile infection (Infections and infestations) | 1 (1)
Device related infection (Infections and infestations) | 1 (1)
Haematoma infection (Infections and infestations) | 1 (1)
Incision site cellulitis (Infections and infestations) | 1 (1)
Klebsiella infection (Infections and infestations) | 1 (1)
Lip infection (Infections and infestations) | 1 (1)
Septic shock (Infections and infestations) | 1 (1)
Vulvovaginal candidiasis (Infections and infestations) | 1 (1)
Wound abcess (Infections and infestations) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 7 (7)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hyperkalaemia (Metabolism and nutrition disorders) | 3 (3)
Fluid overload (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (1)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3 (4)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pyrexia (General disorders) | 5 (5)
Fatigue (General disorders) | 2 (2)
Chills (General disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Oedema peripheral (General disorders) | 1 (1)
Electrocardiogram QT prolonged (Investigations) | 2 (3)
Platelet count decreased (Investigations) | 2 (2)
Blood alkaline phosphatase increased (Investigations) | 1 (1)
Urine output decreased (Investigations) | 1 (1)
Hypotension (Vascular disorders) | 3 (3)
Deep vein thrombosis (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 1 (1)
Haemorrhage (Vascular disorders) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 5 (5)
Tachycardia (Cardiac disorders) | 1 (1)
Anxiety (Psychiatric disorders) | 2 (2)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 1 (1)
Hallucination (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1)
Bladder spasm (Renal and urinary disorders) | 1 (1)
Haematuria (Renal and urinary disorders) | 1 (1)
Pollakiuria (Renal and urinary disorders) | 1 (1)
Urinary retention (Renal and urinary disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (2)
Pruritus generalised (Skin and subcutaneous tissue disorders) | 1 (1)
Skin irritation (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Paraesthesia (Nervous system disorders) | 1 (1)
Presyncope (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 1 (1)
Lacrimation increased (Eye disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No